CLINICAL TRIAL: NCT01701024
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, 2-Arm, Parallel Group Comparison Study Comparing the Efficacy and Safety of ACYC and ACYC Vehicle Gel in the Treatment of Acne Vulgaris
Brief Title: Clinical Study to Test the Efficacy and Safety of ACYC to Treat Moderate to Severe Acne
Acronym: ACYC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V01-ACYC-301
Record Dates: First submitted 2012-09-27; First posted 2012-10-04 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Acne
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACYC (Active Comparator): ACYC active, topically applied to the face for 12 weeks
  Interventions: Drug: ACYC
- ACYC vehicle (Placebo Comparator): ACYC vehicle (placebo), topically applied to the face for 12 weeks
  Interventions: Drug: ACYC vehicle

INTERVENTIONS:
Drug: ACYC — ACYC active, topically applied to the face for 12 weeks
  Arms: ACYC
Drug: ACYC vehicle — ACYC vehicle (placebo), topically applied to the face for 12 weeks
  Arms: ACYC vehicle

SUMMARY:
The primary objective of this study is to compare the efficacy and safety and tolerability of ACYC Gel and vehicle in the treatment of subjects with Acne Vulgaris.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the efficacy and safety and tolerability of ACYC Gel and vehicle in the treatment of subjects with Acne Vulgaris

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female between the ages of 12 and 40 (inclusive)
* Written and verbal informed consent must be obtained.
* Subjects less than 18 years of age must sign an assent for the study and a parent or a legal guardian must sign the informed consent
* Subject must have moderate to severe acne at the baseline visit
* Women of childbearing potential must be willing to practice effective contraception for the duration of the study

Key Exclusion Criteria:

* Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study
* Dermatological conditions on the face that could interfere with clinical evaluations

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 498 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilima Justice, M.D., Study Director — Medical Monitor, Valeant Pharmaceuticals
Locations (24):
- United States (24):
  - Mobile, Alabama
  - Los Angeles, California
  - San Diego, California
  - New Haven, Connecticut
  - Aventura, Florida
  - Naperville, Illinois
  - Evansville, Indiana
  - South Bend, Indiana
  - Louisville, Kentucky
  - Clinton Township, Michigan
  - Fridley, Minnesota
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Rochester, New York
  - Raleigh, North Carolina
  - Portland, Oregon
  - Goodlettsville, Tennessee
  - Austin, Texas
  - College Station, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Lynchburg, Virginia
  - Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACYC | ACYC Vehicle
Started | 253 | 245
Completed | 243 | 236
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACYC | ACYC Vehicle | Total
Number analyzed (Participants) | 253 | 245 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.2 (5.6) | 19.3 (6) | 18.7 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 119 | 242
  Male | 130 | 126 | 256
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 72 | 136
  Not Hispanic or Latino | 189 | 173 | 362
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 33 | 24 | 57
  White | 208 | 210 | 418
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Inflammatory Lesion Count [Mean (Standard Deviation); unit: Lesions] | 27.2 (5.99) | 26.7 (6.09) | 27 (6.04)
Non-Inflammatory Lesion Count [Mean (Standard Deviation); unit: Lesions] | 38.3 (18.63) | 37.2 (17.07) | 37.8 (17.87)
Evaluator's Global Severity Score (EGSS) [Number; unit: participants]
  Clear | 0 | 0 | 0
  Almost Clear | 0 | 0 | 0
  Mild | 0 | 0 | 0
  Moderate | 212 | 200 | 412
  Severe | 41 | 45 | 86
  Very Severe | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Inflammatory Lesion Count
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: Lesion count
Arm/Group | ACYC | ACYC Vehicle
Number analyzed (Participants) | 253 | 245
Lesion count | 16.3 (9.75) | 8.2 (11.55)

2. Primary Outcome: Absolute Change in Non-inflammatory Lesion Count
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | ACYC | ACYC Vehicle
Number analyzed (Participants) | 253 | 245
lesion count | 19.2 (16.18) | 9.6 (17.49)

3. Primary Outcome: Percent of Subjects Who Have a Least a 2 Grade Reduction
Time Frame: Baseline and 12 Weeks
Measure: Number; unit: Percent with >2% reduction
Arm/Group | ACYC | ACYC Vehicle
Number analyzed (Participants) | 253 | 245
Percent with >2% reduction | 35.2 | 17

4. Primary Outcome: Percent of Subjects With Two Grade Reduction From Baseline and Achieving Clear or Almost Clear
Time Frame: Baseline and 12 Weeks
Measure: Number; unit: percentage of clear or almost clear
Arm/Group | ACYC | ACYC Vehicle
Number analyzed (Participants) | 253 | 245
percentage of clear or almost clear | 28.5 | 14.5

ADVERSE EVENTS:
Arm/Group | ACYC | ACYC Vehicle
Serious Adverse Events (participants affected / at risk) | 0/243 | 0/236
Other Adverse Events (participants affected / at risk) | 38/243 | 31/236
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACYC (N=243) | ACYC Vehicle (N=236)
Abdominal Pain (Gastrointestinal disorders) | 0 | 3
Headache (Nervous system disorders) | 3 | 5
Influenza (Infections and infestations) | 5 | 5
Nasopharyngitis (Infections and infestations) | 18 | 12
Pyrexia (General disorders) | 3 | 2
Sinusitis (Infections and infestations) | 7 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No